CLINICAL TRIAL: NCT06404073
Title: RECOVER-ENERGIZE: A Platform Protocol for Evaluation of Interventions for Exercise Intolerance in Post-Acute Sequelae of SARS-CoV-2 Infection (PASC)
Brief Title: RECOVER-ENERGIZE Platform Protocol_Appendix B (Structured Pacing (PEM))
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00112409_B; OT2HL156812 (NIH); NHLBI Grant to RTI (Other Grant/Funding Number: RTI subcontracting with DCRI)
Record Dates: First submitted 2024-05-03; First posted 2024-05-08 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Long COVID; Long Covid19; Long Covid-19
Keywords: PASC; Exercise; PEM (post exertional malaise)
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; Motor Activity

STUDY DESIGN:
Intervention Model Description: This platform protocol is designed to allocate participants into an appropriate intervention appendix based on their symptoms of exercise intolerance or post-exertional malaise (PEM). Once assigned to an appendix, eligible participants are randomized in a 1:1 ratio to either the study intervention group or a control group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Structured Pacing (PEM) (Experimental): Participants in this group will complete weekly pacing sessions for 12 weeks. Pacing sessions will last about 30 minutes, as tolerated. Each participant will meet with a provider 'pacing coach' who has received study-specific education about PEM and how to create and manage pacing strategies for participants. Sessions include PEM symptom and trigger assessment; task, function and activity analysis; adaptations and modifications.
  Interventions: Behavioral: Structured Pacing
- Usual Care (Other): Participants in this group will receive basic education about PEM with a weekly call by site study staff for support and communication.
  Interventions: Other: Usual Care

INTERVENTIONS:
Behavioral: Structured Pacing — Participants in this group will complete weekly pacing sessions for 12 weeks. Pacing sessions will last about 30 minutes, as tolerated. Each participant will meet with a provider 'pacing coach' who has received study-specific education about PEM and how to create and manage pacing strategies for participants. Sessions include PEM symptom and trigger assessment; task, function and activity analysis; adaptations and modifications.
  Arms: Structured Pacing (PEM)
Other: Usual Care — Participants in this group will receive basic education about PEM with a weekly call by site study staff for support and communication.
  Arms: Usual Care

SUMMARY:
This is a platform protocol designed to be flexible so that it is suitable for a range of interventions and settings within diverse health care systems and community settings with incorporation into clinical COVID-19 management programs and treatment plans if results achieve key study outcomes.

This protocol is a prospective, multi-center, multi-arm, randomized, controlled platform trial evaluating interventions to address and improve exercise intolerance and post-exertional malaise (PEM) as manifestations of Post-Acute Sequelae of SARS-CoV-2 Infection (PASC).

The focus of this protocol is to assess interventions that can improve exercise capacity, daily activities tolerance, and quality of life in patients with PASC.

DETAILED DESCRIPTION:
Study interventions will be added to the platform protocol as appendices. Each appendix will leverage all elements of the platform protocol, with additional elements described in the individual appendix. Study intervention appendices may be added or removed according to adaptive design and/or emerging evidence.

The platform protocol enrolls participants who meet study eligibility criteria. After completing initial screening assessments, eligible participants are assigned to one of the study intervention appendices that are actively enrolling. Participants must meet certain criteria within a specific appendix in order to be included in that appendix. Once assigned to an appendix, eligible participants are randomized to either the study intervention group or a control group.

ELIGIBILITY:
• See NCT06404047 for RECOVER-ENERGIZE: Platform Protocol level inclusion and exclusion criteria which applies to this appendix

Additional Appendix B (Structured Pacing (PEM)) Level Inclusion Criteria:

1. Participant identifies new PEM following a SARS-CoV-2 infection that has persisted for at least 12 weeks and is still present at the time of consent
2. Score of 2 or greater for both frequency and severity for any of the first 5 questions on the Screening mDSQ-PEM AND Answer of YES to either item 7 or 8 on Screening mDSQ-PEM, and response of >14 h in item 9.

or Score of 3 or greater on any severity question(regardless) and answer of YES to either item 7 or 8 on the Screening mDSQ-PEM, and response of >14h in item 9.

Additional Appendix B (Structured Pacing (PEM)) Level Exclusion Criteria:

1. Inability to attend in-person screening visit or participate in weekly visits (in-person [≥ 1] and remote)
2. Participant was previously enrolled in Appendix A of this protocol and has NOT completed the full study follow-up period of Appendix A

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2024-07-17 (Actual); Primary Completion 2025-11-17 (Actual); Study Completion 2025-11-17 (Actual)

PRIMARY OUTCOMES:
Change in frequency of PEM symptoms, as measured by the Modified DePaul Symptom - Post-Exertional Malaise questionnaire (mDSQ-PEM) | Baseline, week 12 (End Of Intervention (EOI)), month 6 (End of Study (EOS))
  Symptom frequency is rated on a 5-point Likert scale: 0 = none of the time, 1 = a little of the time, 2 = about half the time, 3 = most of the time, and 4 = all of the time.
Change in severity of PEM symptoms, as measured by the Modified DePaul Symptom - Post-Exertional Malaise questionnaire (mDSQ-PEM) | Baseline, week 12 (EOI), month 6 (EOS)
  Symptom severity is rated on a 5-point Likert scale: 0 = symptom not present, 1 = mild, 2 = moderate, 3 = severe, 4 = very severe.
Change in duration of PEM symptoms, as measured by the Modified DePaul Symptom - Post-Exertional Malaise questionnaire (mDSQ-PEM) | Baseline, week 12 (EOI), month 6 (EOS)

SECONDARY OUTCOMES:
Change in PASC symptoms, as measured by the PASC Symptom Questionnaire | Baseline, week 6 (Middle of Intervention), week 12 (EOI), month 6 (EOS)
  The PASC Symptom Questionnaire is a 33-question survey for self-reporting multiple PASC-related symptoms across multiple systems.
Change in PASC symptoms, as measured by the PROMIS-Cog Questionnaire | Baseline, week 6 (Middle of Intervention), week 12 (EOI), month 6 (EOS)
  The PROMIS Short Form v.2.0 - Cognitive Function 8a (PROMIS-Cog) is the PROMIS Short Form to assess cognitive function and is a self-report, 8-item questionnaire targeting cognitive function in the past seven days.
Change in quality of life, as measured by the PROMIS-29+2 | Baseline, week 6 (Middle of Intervention), week 12 (EOI), month 6 (EOS)
  The PROMIS-29+2 is used to calculate a preference score (PROPr) by the addition of two Cognitive Function Ability items. Preference-based scores provide an overall summary of health-related quality of life on a common metric. Preference-based scores summarize multiple domains on a metric ranging from 0 (as bad as dead) to 1 (perfect or ideal health).
Change in quality of life, as measured by the EQ-5D 5L | Baseline, week 6 (Middle of Intervention), week 12 (EOI), month 6 (EOS)
  The EQ-5D is a standardized measure of health status.
Change in physical activity, as measured by Actigraphy | Baseline, week 6 (Middle of Intervention), week 12 (EOI), month 6 (EOS)
  Actigraphy will be measured by Fitbit.
Change in physical activity, as measured by the PROMIS SF-Physical Function (PROMIS-PF) | Baseline, week 6 (Middle of Intervention), week 12 (EOI), month 6 (EOS)
  The PROMIS Short Form v2.0 - Physical Function 8b (PROMIS-PF) consists of 8 items. The PROMIS Physical Function instruments measure self-reported capability rather than actual performance of physical activities.
Change in orthostatic hypotension, as measured by the Modified Orthostatic Hypotension Questionnaire (mOHQ) | Screening, week 6 (Middle of Intervention), week 12 (EOI), month 6 (EOS)
  The Orthostatic Hypotension Questionnaire (OHQ) is a measure of orthostatic intolerance. The modified OHQ (mOHQ) measure used in this study includes a total of ten items related to daily activities and symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Gary M Felker, MD, Study Chair — Duke Clinical Research Institute; Barry Make, MD, Study Chair — National Jewish Health; Lucinda Bateman, MD, Study Chair — Bateman Horne Center; Janna Friedly, MD, MPH, Study Chair — University of Washington
Locations (1):
- All sites listed under NCT06404047, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
The summary of the results will be shared on the study website: https://recovercovid.org/

REFERENCES:
- See also: Related Info — http://recovercovid.org/

DOCUMENTS (1):
  • Informed Consent Form (2025-04-15): https://cdn.clinicaltrials.gov/large-docs/73/NCT06404073/ICF_000.pdf